CLINICAL TRIAL: NCT06753734
Title: A Cohort Study in Women at High Risk for Gestational Diabetes Based on Breath Metabolomics
Brief Title: Early Prediction of Gestational Diabetes in High-risk Women Based on Breath Metabolomics
Status: Enrolling by invitation | Type: Observational
Sponsor: Tianjin Central Hospital of Gynecology Obstetrics (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KY081
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational Diabetes Group
- control group

SUMMARY:
This study aim to develope novel breath markers of gestational diabetes through a prospective high-risk population cohort study and achieve early prediction of gestational diabetes based on an interpretable machine learning model.

ELIGIBILITY:
Eligibility Criteria

* 18-55 years old
* 11-14 weeks of pregnancy
* at least one risk factor for GDM
* signed a written informed consent

Exclusion Criteria:

* Diabetes mellitus or abnormal glucose metabolism before pregnancy
* Hyperemesis gravidarum (urine ketone positive))
* Thyroid dysfunction
* Asthmatic patients
* Hypertensive diseases that are difficult to control
* Severe hepatic and renal insufficiency or severe electrolyte disturbance
* Malignant tumor
* Acute inflammation
* lung disease
* Patients with gastritis, duodenum and other digestive system diseases
* Those with upper respiratory or oral problems who cannot cooperate with expiratory collection
* smoker

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population in this study include pregnant women aged 18-55 years and at 11-14 weeks gestation with at least one risk factor for GDM
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of gestational diabetes mellitus | 24-28 weeks gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, China